CLINICAL TRIAL: NCT03573752
Title: Study of Outpatient Management for Promontofixation by Laparoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 6796
Record Dates: First submitted 2018-04-05; First posted 2018-06-29 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Pelvic Organ Prolapse
Keywords: Laparoscopic Promontofixation; Outpatient management
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: outpatient management for promontofixation by laparoscopy — postoperative H8 exit after laparoscopic promontofixation
Other: questionnaire — Each patient will complete a questionnaire on the experience of management, both in terms of pain management, anxiety and overall satisfaction.

SUMMARY:
Laparoscopic promontofixation is becoming increasingly common and is currently the standard surgical procedure for pelvic prolapse, with few complications including exposure and mesh infection.

The research hypothesis is that laparoscopic promontofixation is a relatively painless procedure and can be performed on an outpatient basis without increasing the number of postoperative complications and impairing patients' quality of life.

The objective of this study is to evaluate the number of rehospitalizations after management of promontofixation by laparoscopy on an outpatient basis.

To evaluate the feasibility of a postoperative H8 exit after laparoscopic promontofixation.

Each patient will complete a questionnaire on the experience of management, both in terms of pain management, anxiety and overall satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Woman with promontofixation indication by laparoscopy for prolapse cure
* Patient's desire for outpatient management
* Age ≥18 years and <70 years
* Absence of a major medical or surgical history that would prolong hospitalization (ASA 1 or 2, absence of Obstructive Sleep Apnea Syndrome)
* Subject affiliated to a social security scheme
* Subject having signed an informed consent
* Availability of a caregiver, responsible and valid (for the first 48 hours after the potential early exit) at home
* Geographical distance less than one hour from a suitable care facility
* Access to a telephone or a means of transport if necessary
* Patient compliance
* Oral and written comprehension of pre- and post-operative instructions
* Correct housing condition
* Subject having been informed of the results of the prior medical examination

Exclusion Criteria:

* Laparoscopic contraindication
* Comorbidity needs of medical supervision most of 24h
* TVT-O procedure during the same surgery
* Mental handicap affecting autonomy
* Comprehension difficulties to understand the protocol
* No social protection
* Subject with curatorship or guardianship
* Morbid obesity
* Alcohol or drugs addiction
* Excessive anxiety
* Impossibility to give the subject enlightened information (subject in emergency situation...)
* Pregnant woman (positive urinary pregnancy test for women of childbearing age)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Rate of rehospitalizations occurring between outpatient discharge and postoperative follow-up consultation | 35 to 70 Days after the intervention
  Rate of rehospitalizations occurring between outpatient discharge and postoperative

SECONDARY OUTCOMES:
Exit rate at postoperative H8 according to post-anesthesia discharge scoring system score according to Chung. | Hour 8 after the intervention
  This score considers six criteria: vital signs, ambulation, nausea/vomiting, pain, bleeding and voiding. Each criterion is given a score ranging from 0 to 2. Only patients who achieve a score of 9 or more are considered ready for discharge.
Quality of life assessed by the Euroqol EQ-5D index (EuroQol five dimension scale) | Day 0, 3, 7 and 30 after the intervention
  The EQ-5D questionnaire is made up for two components; health state description and evaluation. In description part, health status is measured in terms of five dimensions; mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The respondents self-rate their level of severity for each dimension using three-level (3L) scale; having no problems, having some or moderate problems, being unable to do/having extreme problems. The respondents are asked to choose the statement which best describes their health status of surveyed day.
  In evaluation part, the respondents evaluate their overall health status using the visual analogue scale (EQ-VAS). The patient is asked to mark health status on the day of the interview on a 20 cm vertical scale with end points of 0 and 100. There are notes at the both ends of the scale that the bottom rate (0) corresponds to "the worst health you can imagine", and the highest rate (100) corresponds to "the best health you can imagine".
Assess the satisfaction of the patients by answering a Patient Satisfaction Questionnaire | Day 30 after the intervention
  Assess the satisfaction of the patients by answering a Patient Satisfaction Questionnaire. It includes a satisfaction scale ranging from 0 to 10 and 2 closed-response questions, with the possibility of adding a free comment.
Assess the postoperative anxiety by the State-Trait Anxiety Inventory (STAI) form Y-A. | Day 0, 1, 2, 3, 7 and 30 after the intervention
  Assess the postoperative anxiety by the State-Trait Anxiety Inventory (STAI) form Y-A. This form has 20 items for assessing state anxiety. All items are rated on a 4-point scale. Higher scores indicate greater anxiety.
Assess postoperative pain by the Visual Analogue Scale (VAS) and the consumption of analgesics. | 8 hours after surgery (Day 0)/ At 8 a.m. and 6 p.m. (Day 1, 2 and 3)/ At 8 a.m. (Day 4, 5, 6, 7 and 30)
  Assess postoperative pain by the Visual Analogue Scale (VAS) and the consumption of analgesics. This scale consists of a straight line with the endpoints defining extreme limits such as "no pain at all" and "pain as bad as it could be". The patient is asked to mark his pain level on the line between the two endpoints. The distance between "no pain at all" and the mark then defines the subject's pain.
Rates of postoperative complications | 35 to 70 Days after the intervention
  Rates of postoperative complications
Number of emergency consultations before scheduled postoperative follow-up consultation | 35 to 70 Days after the intervention
  Number of emergency consultations before scheduled postoperative follow-up consultation
Difference in actual costs and cost-effectiveness between conventional and outpatient care | 35 to 70 Days after the intervention
  Collection of the PMSI (medical information system program) of the made act and the cost of the hospital stay in ambulatory for a laparoscopic promontofixation.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de gynécologie, Centre Médico Chirurgical Obstétrical, Hôpitaux Universitaires de Strasbourg, Schiltigheim, France

REFERENCES:
- [Result] Collin-Bund V, Viviani V, Meyer N, Goetsch T, Boisrame T, Faller E, Lecointre L, Gabriele V, Akladios C, Garbin O, Host A. Study of the feasibility of outpatient sacrocolpopexy by laparoscopy. J Gynecol Obstet Hum Reprod. 2024 Sep;53(7):102792. doi: 10.1016/j.jogoh.2024.102792. Epub 2024 Apr 23. PMID 38663686